CLINICAL TRIAL: NCT00994812
Title: Effects of Metformin on Fertility and Pregnancy in Women With Polycystic Ovary Syndrome: a Randomized, Prospective, Placebo-controlled Multicenter Study
Brief Title: The Effects of Metformin on Pregnancy and Miscarriage Rates in Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: University of Eastern Finland (Other); University of Helsinki (Other); Tampere University (Other); University of Turku (Other)
Responsible Party: Laure Morin-Papunen/ Associate Professor, Dept of Obstetrics and Gynecology, University Hospital of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T59108
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2009-10

CONDITIONS: Polycystic Ovary Syndrome; Miscarriage; Infertility; Toxemia; Gestational Diabetes
Keywords: Polycystic ovary syndrome; PCOS; Metformin; Miscarriage; Infertility; Complications of pregnancy
MeSH Terms: conditions — Polycystic Ovary Syndrome; Abortion, Spontaneous; Infertility; Toxemia; Diabetes, Gestational; Pregnancy Complications | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin — The obese women will be randomized either to metformin (2g/day) or to placebo, and the non-obese either to metformin (1.5g/day) or to placebo. All subjects will be evaluated 1 to 7 days after spontaneous menstruation (oligomenorrheic patients), or at any other convenient time (amenorrheic subjects). After the treatment of 3 months with metformin/placebo alone, another appropriate infertility treatment will be combined with metformin/placebo (clomiphene, ovulation induction, insemination or in vitro fertilization) if no pregnancy has occurred. This treatment will be continued another 6 months' period. If pregnancy occurs, subjects will be re-examined at 7-8 weeks of gestation.

SUMMARY:
The purpose of this study is to determine whether metformin may improve pregnancy rates, and decrease miscarriage rates and complications of pregnancy, such as toxemia and gestational diabetes, in women with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Women with PCOS represent about 5-10% of the general female population and one third of the women treated for infertility. Thus, the development of new therapies to improve the efficiency of ovulation induction treatments and the outcome of pregnancy, and to reduce the long-term risks of the syndrome would bring important health benefits.

The central role played by insulin resistance and hyperinsulinemia in PCOS - causing hyperandrogenism, premature follicular atresia, anovulation, oligo-amenorrhea and anovulatory infertility - has led to the use of insulin-lowering drugs for the treatment of this syndrome. The most studied agent is metformin, a biguanide antihyperglycemic drug used to treat Type 2 diabetes mellitus. It has been shown to improve significantly hyperinsulinemia and insulin resistance, to decrease androgen levels, and to improve menstrual pattern and, alone or in addition to clomiphene citrate, to induce ovulation and improve pregnancy rates in women with PCOS in some studies (1,2). Metformin may also decrease risks of early spontaneous miscarriage and gestational diabetes in PCOS (3-6). Two recent RCTs, however, have shown no beneficial effect of metformin compared to placebo as regards rates of pregnancy, miscarriage or life births in women with PCOS (7,8).

Our hypothesis is that metformin may improve pregnancy rates and decrease miscarriage occurrence and complications of pregnancy, such as toxemia and gestational diabetes, in women with PCOS. This multicenter randomized placebo-controlled study is conducted in all five University Hospitals of Finland (Oulu, Kuopio, Helsinki, Tampere and Turku). Blood samples are drawn and the oral glucose tolerance test (OGTT) done before and at 3 months of treatment, after which the treatment with placebo/metformin is continued another 6 months' period together with the appropriate infertility treatment. If pregnancy occurs, the OGTT is done at 7-8 weeks of pregnancy and the placebo/metformin treatment is continued until 12 weeks of pregnancy. The study has already started and is estimated to continue at least until the end of 2009. Power analysis indicated that a minimum of 60 pregnant patients are needed in each group to decrease the risk of miscarriage from 44% to the normal 15%.

ELIGIBILITY:
Inclusion Criteria:

1. age < 40 years at entry
2. BMI > 19 kg/m2
3. Infertility lasting > 1 year
4. Criteria for PCOS are as defined by ESHRE/ASRM: at least two of the following findings:

   * polycystic ovaries shown by vaginal ultrasonography (more than 12 subcapsular follicles of 3-8 mm diameter in one plane of the ovary)
   * oligomenorrhea or amenorrhea
   * clinical manifestations of hyperandrogenism such as a hirsutism score of > 7 according to Ferriman and Gallwey (Ferriman & Gallwey 1961)and/or an elevated serum testosterone level (> 2.7 nmol/l).

Exclusion Criteria:

1. diabetic subjects
2. alcohol users
3. active liver disease (ALAT > +2 SD the upper normal value i.e.> 100IU/l)
4. hormonal drugs
5. past or present cardiac failure (NYHA I-IV)
6. liver or renal failure (S-Creatinine above the normal value ie.124 umol/l)
7. pregnancy or lactation
8. hypersensitivity to metformin

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2002-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Miscarriage rates | at 7-8 weeks of pregnancy or later if miscarriage happens later

SECONDARY OUTCOMES:
Effect of metformin versus placebo on the time to be pregnant | 3-6 months
Effect of metformin versus placebo on the rates of toxemia during pregnancy | 3 months after birth of the child
Effects of metformin versus placebo on the rates of gestational diabetes during pregnancy | 3 months after the birth of the child

CONTACTS AND LOCATIONS:
Overall Officials: Laure C Morin-Papunen, PhD, Principal Investigator — University hospital of Oulu
Locations (5):
- Finland (5):
  - University Hospital Of Helsinki, Helsinki
  - University Hospital of Kuopio, Kuopio
  - University Hopsital of Oulu, Oulu
  - University Hospital of Tampere, Tampere
  - University Hospital of Turku, Turku

REFERENCES:
- [Background] Kashyap S, Wells GA, Rosenwaks Z. Insulin-sensitizing agents as primary therapy for patients with polycystic ovarian syndrome. Hum Reprod. 2004 Nov;19(11):2474-83. doi: 10.1093/humrep/deh440. Epub 2004 Sep 9. PMID 15358717
- [Background] Glueck CJ, Phillips H, Cameron D, Sieve-Smith L, Wang P. Continuing metformin throughout pregnancy in women with polycystic ovary syndrome appears to safely reduce first-trimester spontaneous abortion: a pilot study. Fertil Steril. 2001 Jan;75(1):46-52. doi: 10.1016/s0015-0282(00)01666-6. PMID 11163815
- [Background] Glueck CJ, Wang P, Kobayashi S, Phillips H, Sieve-Smith L. Metformin therapy throughout pregnancy reduces the development of gestational diabetes in women with polycystic ovary syndrome. Fertil Steril. 2002 Mar;77(3):520-5. doi: 10.1016/s0015-0282(01)03202-2. PMID 11872206
- [Background] Jakubowicz DJ, Iuorno MJ, Jakubowicz S, Roberts KA, Nestler JE. Effects of metformin on early pregnancy loss in the polycystic ovary syndrome. J Clin Endocrinol Metab. 2002 Feb;87(2):524-9. doi: 10.1210/jcem.87.2.8207. PMID 11836280
- [Background] Palomba S, Orio F Jr, Falbo A, Manguso F, Russo T, Cascella T, Tolino A, Carmina E, Colao A, Zullo F. Prospective parallel randomized, double-blind, double-dummy controlled clinical trial comparing clomiphene citrate and metformin as the first-line treatment for ovulation induction in nonobese anovulatory women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Jul;90(7):4068-74. doi: 10.1210/jc.2005-0110. Epub 2005 Apr 19. PMID 15840746
- [Background] Legro RS, Barnhart HX, Schlaff WD, Carr BR, Diamond MP, Carson SA, Steinkampf MP, Coutifaris C, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Giudice LC, Leppert PC, Myers ER; Cooperative Multicenter Reproductive Medicine Network. Clomiphene, metformin, or both for infertility in the polycystic ovary syndrome. N Engl J Med. 2007 Feb 8;356(6):551-66. doi: 10.1056/NEJMoa063971. PMID 17287476
- [Background] Moll E, Bossuyt PM, Korevaar JC, Lambalk CB, van der Veen F. Effect of clomifene citrate plus metformin and clomifene citrate plus placebo on induction of ovulation in women with newly diagnosed polycystic ovary syndrome: randomised double blind clinical trial. BMJ. 2006 Jun 24;332(7556):1485. doi: 10.1136/bmj.38867.631551.55. Epub 2006 Jun 12. PMID 16769748
- [Derived] Lingaiah S, Morin-Papunen L, Risteli J, Tapanainen JS. Metformin decreases bone turnover markers in polycystic ovary syndrome: a post hoc study. Fertil Steril. 2019 Aug;112(2):362-370. doi: 10.1016/j.fertnstert.2019.04.013. Epub 2019 Jun 18. PMID 31227287
- [Derived] Sova H, Puistola U, Morin-Papunen L, Karihtala P. Metformin decreases serum 8-hydroxy-2'-deoxyguanosine levels in polycystic ovary syndrome. Fertil Steril. 2013 Feb;99(2):593-8. doi: 10.1016/j.fertnstert.2012.10.013. Epub 2012 Oct 31. PMID 23122829